CLINICAL TRIAL: NCT06834633
Title: Impact of a Nephroprotection Bundle-of-care in Severe Trauma Patients at Risk of Acute Kidney Injury: a Multicenter Randomized Controlled Trial
Brief Title: Nephroprotection in Severe Trauma Patients With Kidney Stress
Acronym: NephroTrauma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL21_1435; 2022-A01052-41 (Other: ID-RCB)
Record Dates: First submitted 2024-11-04; First posted 2025-02-19 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Trauma; Complications
Keywords: Severe trauma; Acute Kidney Injury; Nephroprotection bundle-of-care; Biomarker
MeSH Terms: conditions — Wounds and Injuries; Acute Kidney Injury | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The study will be conducted in two phases:
  Observational phase (4 months): describe the usual management practices and the incidence of AKI in each center.
  Severe trauma patients (ISS >15) will have a urine sample taken for NC measurement within 12 hours of admission to critical care. The NC value will not be disclosed to practitioners. Only patients with NC>0.3 will be included retrospectively Interventional phase (20 months): aims to evaluate the effectiveness of a nephroprotection bundle-of-care (adaptation of the "KDIGO" protocol).
  Patients with ISS>15 will have a urine sample taken for NC measurement within 12 hours of admission to critical care. The NC result will be returned to the practitioner. If NC > 0.3, the patient can be included and randomized. Randomization will be stratified by center. In the intervention group, the nephroprotection bundle-of-care will be applied for 3 days following admission to critical care. In the control group, patients will be managed as usual
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Observational group (Other): Patients in the observational group will be managed according to the unit's standard-of-care, as in the control group, but without investigators knowing the patient's risk of AKI (NC score not known)
  Interventions: Other: Standard-of-care
- Control group: Standard-of-care (Other): Patients at risk of AKI (NC>0.3) randomized in the control group will be managed according to the unit's standard-of-care.
  Interventions: Other: Standard-of-care
- Intervention group: nephroprotection bundle-of-care (Experimental): Patients at risk of AKI (NC>0.3) randomized in the intervention group will receive the systematic and complete application of a nephroprotection bundle-of-care for three days following ICU admission.
  Interventions: Other: Systematic nephroprotection bundle-of-care

INTERVENTIONS:
Other: Standard-of-care — Management according to current ICU practices
  Arms: Control group: Standard-of-care; Observational group
Other: Systematic nephroprotection bundle-of-care — The nephroprotection bundle-of-care includes 5 components:
  1. Prevention of drugs' nephrotoxicity
  2. Hemodynamic optimization, for 24h
  3. Blood glucose control and avoidance of hyperglycemia
  4. Early detection of rhabdomyolysis
  5. Monitoring of renal function
  Arms: Intervention group: nephroprotection bundle-of-care

SUMMARY:
Acute Kidney Injury (AKI) occurs in 24% of trauma patients, and is even more common in those with severe trauma. It is a major contributor to morbidity and mortality in trauma. Diagnosis of AKI is based on elevated serum creatinine and decreased urine output, two functional markers already indicating the presence of a significant kidney function impairment. Earlier detection of kidney stress, at a preclinical stage when cellular modifications are still reversible, could reduce the occurrence of AKI episodes if nephroprotective measures are rapidly implemented.

Several randomized controlled trials have shown that early implementation of such a nephroprotection bundle-of-care in patients at risk of AKI after major surgery reduces the incidence of severe AKI within 72 hours. Although its use is supported by international guidelines, this nephroprotection bundle-of-care is rarely implemented in its totality, due to the significant financial and human resources required for its full implementation.

The Nephrocheck® (NC) test is a urine test for which a result > 0.3 is predictive of AKI development. It might enable early identification of trauma patients at risk of AKI, so that implementation of the nephroprotection bundle-of-care could be targeted solely at those high-risk patients.

Thus, the investigators hypothesize that in a population of severe trauma patients (ISS score>15) at risk of AKI (defined by a NC on Intensive Care Unit (ICU) admission > 0.3), early implementation of a nephroprotection bundle-of-care would reduce the risk of AKI occurring within 3 days of ICU admission, compared with standard-of-care management. This study will compare the occurrence of AKI in these two groups in a multicenter randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years)
* Severe trauma patients (ISS score > 15) admitted to a trauma center
* Time between trauma and admission to trauma center <6h
* Patient with indwelling urinary catheter
* High risk of AKI: measurement of NC score on fresh urine performed as soon as possible within 12 hours of admission to ICU and value > 0.3.
* Affiliated with a social security scheme or beneficiary of a similar scheme
* Consent signed by patient or close relative, or attestation signed by investigator in case of emergency

Exclusion Criteria:

* Adult under legal protection (guardianship, curators)
* Persons deprived of their liberty by judicial or administrative decision
* Patients taking part in other interventional research which may interfere with the research and which includes an exclusion period still in progress at the time of inclusion.
* Pregnant or breast-feeding woman (diagnosis of pregnancy by plasma βHCG (Beta-Human Chorionic Gonadotropin) assay routinely performed as part of the blood test on admission to the outpatient department of a woman of childbearing age).
* Patients with end-stage or severe chronic renal failure with Glomerular Filtration Rate (GFR) < 30 milliliters/min/1.73m2 or chronic dialysis.
* Anuric patients
* Severe heart failure defined as Left Ventricular Ejection Fraction (LVEF) <25%.
* Patient moribund on admission with an estimated length of stay of less than 24 hours
* Patient with AKI at time of randomization (developed prior to ICU admission or within the first 12 hours of ICU admission, before randomization).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 523 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients developing an AKI episode within 3 days after ICU admission. | During 3 days from ICU admission.
  AKI will be defined according to KDIGO (Kidney Disease: Improving Global Outcomes) criteria, either by a drop in urine output (oliguria < 0.5ml/kg/h for 6h) and/or a rise in serum creatinine (1.5x baseline or increase of 26.5 µmol/l).

SECONDARY OUTCOMES:
Proportion of patients with AKI within 7 days of ICU admission | During 7 days from ICU admission
  AKI will be defined according to KDIGO criteria, either by a drop in urine output (oliguria < 0.5ml/kg/h for 6h) and/or a rise in serum creatinine (1.5x baseline or increase of 26.5 µmol/l).
Proportion of patients with severe AKI within 3 days of ICU admission | During 3 days from ICU admission
  Severe AKI is defined as AKI stage 2 or 3 according to KDIGO criteria
Proportion of patients with severe AKI within 7 days of ICU admission | During 7 days from ICU admission
  Severe AKI is defined as AKI stage 2 or 3 according to KDIGO criteria
Proportion of patients with MAKE (MAjor Adverse Kidney Event) 28 | At 28 days after ICU admission
  MAKE 28 is defined by the occurrence of one event among (1) death before day 28 after ICU admission, (2) requirement of renal replacement therapy on day 28 or (3) incomplete renal recovery on day 28.
Proportion of patients with a complication among cardiovascular and hemodynamic complications; septic complications; hemorrhagic complications within 7 days after ICU admission | During 7 days after ICU admission.
  Cardiovascular or hemodynamic complications include ventricular cardiac rhythm disorders, cardiogenic acute pulmonary edema and poorly controlled arterial hypertension [MAP (Mean Arterial Pressure) > 120 mmHg for 4 hours].
  Septic complications correspond to sepsis defined by the association of an infection and an increase in SOFA >=2.
  Hemorrhagic complications are defined by the number of packed red blood cells (RBCs) used.
Proportion of patients with at least one episode of dysglycemia within 3 days after ICU admission | During 3 days after ICU admission.
  Episodes of dysglycemia are defined as hypoglycemia (<4mmol/l) or hyperglycemia (>12mmol/l).
ICU and hospital length-of-stay | During 28 days from ICU admission
  Total number of days spent in critical care (intensive care, continuous care) and in the initial hospital
Identification of risk factors for AKI in trauma patients using clinical and laboratory parameters | During 7 days from ICU admission
  Known and novel risk factors for AKI in trauma patients will be evaluated using clinical variables (e.g., age, comorbidities, injury severity scores), hemodynamic parameters (e.g., MAP, lactate), and biomarkers of kidney function (e.g., CPK, TIMP-2/IGFBP-7)
Incidence of AKI in trauma patients within 3 days of ICU admission based on KDIGO Criteria | During 3 days after ICU admission
  The incidence of all stages and severe AKI in trauma patients at risk will be assessed based on the KDIGO criteria
Characterization of AKI episodes phenotype in trauma patients using KDIGO criteria | During 7 days from ICU admission
  Acute Kidney Injury episodes will be characterized based on a combination of factors including :
  * Time to AKI onset: defined as the time (in hours) from ICU admission to the diagnosis of AKI
  * Diagnostic criteria: whether the AKI is diagnosed based on serum creatinine or urine output changes
  * Severity: the highest KDIGO stage (1, 2, or 3) reached during the episode
  * Duration: transient (<48h) or persistent (≥48h) AKI.
Proportion of patients receiving the nephroprotection bundle-of-care in its entirety, by component, and by practice. | During 3 days after ICU admission
  The entirety of the nephroprotection bundle-of-care is defined by the combination of at least one practice from each component: medication, hemodynamics, rhabdomyolysis, monitoring, glycemia
Cost-effectiveness incremental ratio of the nephroprotection bundle-of-care compared with standard-of-care at 7 days after ICU admission. | At 7 days after ICU admission
  The incremental cost-effectiveness ratio will be expressed as the additional cost per AKI avoided.
Cost-effectiveness incremental ratio of the nephroprotection bundle-of-care compared with standard-of-care at 28 days after ICU admission. | At 28 days after ICU admission
  The incremental cost-effectiveness ratio will be expressed as the additional cost per AKI avoided.
Average costs of initial hospital stay for each group | During 28 days after ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Céline MONARD, Principal Investigator — Hospices Civils de Lyon
Locations (6):
- France (6):
  - Centre Hospitalier universitaire Estaing, Service anesthésie-réanimation, Clermont-Ferrand
  - Centre hospitaler Annecy Genevois, Service de réanimation, Épagny
  - Centre hospitalier universitaire de Grenoble Alpes, Pôle anesthésie-réanimation, La Tronche
  - Hospices Civils de Lyon, Hôpital Edouard Herriot, Service d'anesthésie-réanimation, Lyon
  - Hospices Civils de Lyon, Hôpital Lyon-Sud, Service d'anesthésie-réanimation, Pierre-Bénite
  - Centre hospitalier universitaire de Saint Etienne, Hôpital Bellevue, Service anesthésie-réanimation, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No